CLINICAL TRIAL: NCT05673187
Title: A Multicentre, Single-arm Phase II Trial of Adagrasib in Patients With KRASG12C-mutant NSCLC, Including the Elderly (≥70 Years) or Patients With Poor Performance Status
Brief Title: Adagrasib in Patients With KRASG12C-mutant NSCLC Who Are Elderly or Have Poor Performance Status
Acronym: ADEPPT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 22-22; 2022-002736-31 (EudraCT Number)
Record Dates: First submitted 2022-11-14; First posted 2023-01-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: NSCLC Stage IV; KRAS P.G12C
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — adagrasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Adagrasib to be administered at a dose of 600 mg orally, twice daily until progression or unacceptable toxicity.
  Interventions: Drug: Adagrasib

INTERVENTIONS:
Drug: Adagrasib — Adagrasib is administered at a dose of 600 mg orally, twice daily until progression or unacceptable toxicity.

SUMMARY:
ADEPPT is an international, multicentre, single-arm phase II trial. The protocol treatment consists of adagrasib, which is administered at a dose of 600 mg orally, twice daily until progression or unacceptable toxicity.The primary objective of this trial is to assess the clinical efficacy of adagrasib treatment, in terms of objective response, in patients with KRASG12C-mutant NSCLC, including the elderly (≥70 years) or patients with poor performance status (ECOG PS=2).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed stage IV NSCLC.
2. KRASG12C-mutation by local testing (by tissue or ctDNA).
3. Prior treatment with at least one line of systemic therapy for NSCLC (e.g., platinum-based doublet chemotherapy and/or immune-checkpoint inhibition or both).
4. Life expectancy ≥12 weeks.
5. Measurable disease according to RECIST v1.1.
6. Age ≥18 years with ECOG PS 2 (cohort 1), or age ≥70 years with ECOG PS 0-1 (cohort 2).
7. Adequate haematological, renal and liver function
8. Men and women of childbearing potential must agree to use use highly effective contraceptive methods.
9. Women of childbearing potential, including women who had their last menstruation in the last 2 years, must have a negative urinary or serum beta HCG pregnancy test within 5 weeks before enrolment. Pregnancy test must be repeated within 7 days before the first dose of adagrasib treatment.Ability to comply with the trial protocol, in the investigator's judgment.
10. Written IC for study participation must be signed and dated by the patient and the investigator prior to any study-related intervention, including the submission of mandatory biomaterial.

Exclusion Criteria:

1. Prior investigational therapy within 28 days or at least 5 half-lives before enrolment.
2. Prior treatment with an agent targeting KRASG12C.
3. Leptomeningeal disease or untreated brain metastases.

   * Patient should be neurologically stable for at least 2 weeks before enrolment, without the need for corticosteroids, except for prednisone (or its equivalent) at a dose of ≤10 mg daily.
   * For patients with definitively treated brain metastases, a time period of minimum of 2 weeks must have elapsed from the last day of radiotherapy.
4. History of intestinal disease or major gastric surgery likely to alter absorption of study treatment or inability to swallow oral medications.
5. Any of the following cardiac abnormalities:

   * Unstable angina pectoris or myocardial infarction within 6 months prior to enrolment.
   * Symptomatic or uncontrolled atrial fibrillation within 6 months prior to enrolment.
   * Congestive heart failure ≥NYHA Class 3 within 6 months prior to enrolment.
   * Prolonged QTc interval >480 ms or family or medical history of congenital Long QT Syndrome.
6. History of stroke or transient ischemic attack within 6 months prior to enrolment.
7. Ongoing need for treatment with concomitant medication with any of the following characteristics: known risk of Torsades de Pointes; substrate of CYP3A with narrow therapeutic index; strong inducer of CYP3A and/or P-gp; strong inhibitor of BCRP; and proton pump inhibitors that cannot be switched to alternative treatment prior to enrolment.
8. Known human immunodeficiency virus (HIV) infection.
9. Acute or chronic hepatitis B or C infection.
10. Women who are pregnant or in the period of lactation.
11. Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the study.
12. Judgement by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per RECIST v1.1, assessed at 12 weeks. | From date of enrolment until 12 weeks post-enrolment
  The primary objective of this trial is to assess the clinical efficacy of adagrasib treatment, in terms of objective response as defined as the rate of patients achieving a best overall response [complete response (CR) or partial response (PR)] according to RECIST v1.1

SECONDARY OUTCOMES:
Durable clinical benefit | From date of enrolment until at least the 24-week assessment.
  Durable clinical benefit (DCB) is defined as the rate among all enrolled patients who are alive and without disease progression who achieve CR or PR, according to RECIST v1.1, or stable disease (SD) lasting for at least 24 weeks.
Time-to-progression (TTP) | From the date of enrolment until last tumour assessment (approximately 20-26 months after enrolment of the first patient)
  Time-to-progression (TTP) is defined as the time from the date of enrolment until the date of documented progression (according to RECIST v1.1). Censoring for patients without documented progression will occur at the date of last tumour assessment without PD. Patients without a post-baseline tumour assessment will be censored at the date of enrolment plus 1 day.
Progression-free survival (PFS) | From the date of enrolment until last tumour assessment (approximately 20-26 months after enrolment of the first patient)
  Progression-free survival (PFS) is defined as the time from the date of enrolment until the date of documented progression (according to RECIST v1.1) or death, if progression is not documented. Censoring (for patients without progression or death) will occur at the date of last tumour assessment. Patients without a post-baseline tumour assessment will be censored at the date of enrolment plus 1 day.
Overall survival (OS) | From the date of enrolment until last patient last visit (approximately 20-26 months after enrolment of the first patient)
  Overall survival (OS) is defined as the time from the date of enrolment until the date of death from any cause. Censoring for patients who are not reported as dead will occur at the last date they are known to be alive. Data for patients who do not have post-baseline information will be censored at the date of enrolment plus 1 day.
Safety and tolerability | From the date of enrolment until last patient last visit (approximately 20-26 months after enrolment of the first patient)
  The toxicity and safety profile of the protocol treatment will be evaluated by:
  * Adverse events (AEs) according to CTCAE v5.0 (any-cause, as well as treatment-related) including AEs leading to dose delays and/or interruptions, withdrawal of protocol treatment, and death
  * Severe and serious AEs
  * Deaths
Laboratory parameters and abnormalities 1 | From the date of enrolment until last patient last visit (approximately 20-26 months after enrolment of the first patient)
  Hemoglobin [g/dl]
Laboratory parameters and abnormalities 2 | From the date of enrolment until last patient last visit (approximately 20-26 months after enrolment of the first patient)
  Platelet count [G/L]
Laboratory parameters and abnormalities 3 | From the date of enrolment until last patient last visit (approximately 20-26 months after enrolment of the first patient)
  White blood cell count [G/L]
Vital signs 1 | From the date of enrolment until last patient last visit (approximately 20-26 months after enrolment of the first patient)
  Blood pressure systolic [mmHg]
Vital signs 2 | From the date of enrolment until last patient last visit (approximately 20-26 months after enrolment of the first patient)
  Blood pressure diastolic [mmHG]
Vital signs 3 | From the date of enrolment until last patient last visit (approximately 20-26 months after enrolment of the first patient)
  Heart rate [beats/min]
Vital signs 4 | From the date of enrolment until last patient last visit (approximately 20-26 months after enrolment of the first patient)
  Body temperature [°C]
Patient-reported outcomes NFLSI-17 | From the date of screening until patient's end of treatment (approximately 20-26 months after enrolment of the first patient)
  Patient-reported symptoms and functioning will be assessed by NCCN-Functional Assessment of Cancer Therapy (FACT) Lung Symptom Index-17 (NFLSI-17).
Patient-reported outcomes PRO-CTCAE® | From the date of screening until patient's end of treatment (approximately 20-26 months after enrolment of the first patient)
  The most commonly reported treatment-related adverse effects of adagrasib (diarrhoea and vomiting) that are not covered by the NFLSI-17 will be assessed by the NCI Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE®).

CONTACTS AND LOCATIONS:
Overall Officials: Jarushka Naidoo, Study Chair — Beaumont RCSI Cancer Centre, Beaumont Hospital
Locations (22):
- Instiute Jules Bordet, Brussels, Belgium
- France (4):
  - Centre Hospitalier d'Avignon, Avignon
  - Caen - CHU, Caen
  - Le Mans - CHG, Le Mans
  - Hôpital de Marseille, Marseille
- Ireland (4):
  - Beaumont Hospital, Dublin
  - St James's Hospital, Dublin
  - University Hospital Limerick, Limerick
  - University Hospital Waterford, Waterford
- Italy (4):
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Santa Maria della Misericordia Hospital, Perugia
  - Istituto Nazionale Tumori "Regina Elena", Rome
  - AULSS2 Marca Trevigiana Treviso, Treviso
- Spain (8):
  - Complejo Hospitalario Universitario a Coruña, A Coruña
  - Alicante University Hospital, Alicante
  - ICO Badalona - Hospital Germans Trias i Pujol, Badalona
  - Hospital de Basurto, Bilbao
  - ICO Bellvitge -H. Duran i Reynals / H. Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital General Universitario de Valencia (University Hospital Valencia), Valencia
- Christie NHS Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP